CLINICAL TRIAL: NCT05493046
Title: Effects of Interactive Hand Exercise Game on Grip Strength and Vascular Maturation in Patients Undergoing Arteriovenous Fistula Surgery: A Randomized Controlled Trial
Brief Title: Interactive Hand Exercise Game on Grip Strength and Vascular Maturation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Collaborators: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Hsiao-Yean Chiu, Associate Professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 22MMHIS083e
Record Dates: First submitted 2022-08-04; First posted 2022-08-09 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Muscle Weakness; Angiogenesis
Keywords: Hand-grip Strength; Hemodialysis
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will be unaware of the treatment assignment before the completion of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interactive Hand Exercise Game (Experimental): Participants will receive an Interactive Hand Exercise Game for 30 minutes every day for consecutive two months.
  Interventions: Behavioral: Interactive Hand Exercise Game
- Soft ball exercise ( routine care) (Active Comparator): Participants will receive a soft ball exercise for 30 minutes every day for consecutive two months.
  Interventions: Behavioral: Soft ball exercise ( routine care)

INTERVENTIONS:
Behavioral: Interactive Hand Exercise Game — Interactive Hand Exercise Game to Improve Vascular Maturity and Grip Strength in Patients undergoing Arteriovenous Fistula Surgery
  Arms: Interactive Hand Exercise Game
Behavioral: Soft ball exercise ( routine care) — Soft ball exercise ( routine care)
  Arms: Soft ball exercise ( routine care)

SUMMARY:
Hemodialysis is currently the most commonly used renal replacement therapy. Compared with arteriovenous graft, central venous catheter, and autologous arteriovenous fistula, the possibility of postoperative re-dredging is low and there are few complications, so isometric hand exercise training is the first choice for hemodialysis strategy.

The intervention of smart technology has greatly improved the treatment effect and quality of life of patients, and it has unique advantages when applied to health care or behavior change intervention programs. This study expects to enhance hand grip strength through interactive hand exercise games combined with grip strength equipment, thereby increasing the vascular maturity of patients with postoperative autologous arteriovenous fistula, and enhancing the motivation of patients to participate.

DETAILED DESCRIPTION:
Hemodialysis is currently the most commonly used renal replacement therapy. Compared with arteriovenous graft, central venous catheter, and autologous arteriovenous fistula, the possibility of postoperative re-dredging is low and there are few complications, so isometric hand exercise training is the first choice for hemodialysis strategy.

The intervention of smart technology has greatly improved the treatment effect and quality of life of patients, and it has unique advantages when applied to health care or behavior change intervention programs. This study expects to enhance hand grip strength through interactive hand exercise games combined with grip strength equipment, thereby increasing the vascular maturity of patients with a postoperative autologous arteriovenous fistula, and enhancing the motivation of patients to participate.

The patients will be assigned to the experimental group and the control group by a simple random method, with 15 patients in each group. The experimental group was guided by the interactive hand exercise game program, while the control group received conventional softball exercise. Two groups of patients will start to perform hand exercises on the first day after returning home. The two groups need to perform 30 minutes each time, twice a day (once in the morning and once in the afternoon), for a total of two months. To assess the study outcomes (i.e., hand grip strength and maturation) will use self-structured questionnaires, Noblus ultrasonic machine and Jamar hydraulic grip. The measurement time points are the one week before, the first week, the fourth weeks and the eighth weeks after the autologous arteriovenous fistula operation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic renal failure stage 4 to 5 (before dialysis) and stage 5 (patients who have started hemodialysis).
* Newly established surgical patients with autologous arteriovenous fistula.
* Aged between 20 and 70 years old.
* Having clear consciousness and being able to communicate in Chinese.

Exclusion Criteria:

* Previous dysfunction of an autologous arteriovenous fistula in the same arm.
* Injury to the fistula extremity.
* Neuromusculoskeletal abnormalities.
* Upper extremity arthritis.
* Peripheral neuropathy.
* Peripheral arterial dysfunction.
* Venous disease.
* Rheumatic disease.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Changes in vein diameter | The 1th week, the 4th weeks and the 8th weeks after the autologous arteriovenous fistula surgery
  This will be measured by using duplex ultrasound. The maturation of autologous arteriovenous fistula is defined as a cross-sectional luminal diameter of the draining vein >6 mm.
Changes in the depth of the fistula from the epidermis | The 1th week, the 4th weeks and the 8th weeks after the autologous arteriovenous fistula operation.
  The depth of the fistula from the epidermis is measured using duplex ultrasound. The maturation of autologous arteriovenous fistula should be <0.6 cm from the epidermis.
Changes in brachial artery blood flow rate | The 1th week, the 4th weeks and the 8th weeks after the autologous arteriovenous fistula operation.
  The flow rate is measured using duplex ultrasound. The maturation of autologous arteriovenous fistula is defined as a flow velocity in the artery >600 ml/min.

SECONDARY OUTCOMES:
Changes in grip strength | The 1th week, the 4th weeks and the 8th weeks after the autologous arteriovenous fistula operation.
  The grip strength is measured using the Jamar Grip. The size is set to 2 for women, 1 for those with smaller hands, and 3 for men.

CONTACTS AND LOCATIONS:
Overall Officials: Chiu Hsiao-Yean, PhD, Principal Investigator — Taipei Medical University
Locations (1):
- Hsiao-Yean Chiu, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luo YC, Han PH, Chen YY, Wu PC, Wu IW, Fan YC, Chiu HY. Effects of Interactive Handgrip Game on Vascular Maturation and Grip Strength in Patients Undergoing Arteriovenous Fistula Surgery: A Feasibility Randomized Controlled Trial. Hemodial Int. 2026 Jan 1. doi: 10.1111/hdi.70045. Online ahead of print. PMID 41479242